CLINICAL TRIAL: NCT01885988
Title: Nebivolol Effects on Endothelial Function and Erectile Function in Non-smoking Pre-hypertensive and Newly Diagnosed Stage 1 Hypertensive Men With Erectile Dysfunction.
Brief Title: Nebivolol Effects on Endothelial Function and Erectile Function
Acronym: NEB-ED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin M. Miner, MD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Martin M. Miner, MD, Co-Director Men's Health Center, The Miriam Hospital
Organization: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BYS-IT-74
Record Dates: First submitted 2013-06-14; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Nebivolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol 5, 10 or 20 mg tablet, oral, daily for 3 months. Nebivolol dosage will be titrated per blood pressure results.
  Interventions: Drug: Nebivolol
- Sugar pill (Placebo Comparator): Sugar pill 5, 10 or 20 mg tablet, orally, daily. Sugar pill dosage will be titrated per blood pressure results.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 5, 10 or 20 mg tablet, oral, daily for 3 months. Nebivolol dosage will be titrated per blood pressure results.
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Sugar Pill — Sugar pill 5, 10 or 20mg taken by mouth, daily. Sugar pill dosage will be titrated per blood pressure results.
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
The study will take part at The Men's Health Center It will involve men who have a diagnosis of erectile dysfunction and also have high blood pressure.

High blood pressure can affect the lining of the arteries and cause stiffness in the arteries. The arteries and veins throughout the body have a lining called the endothelium which gives them the ability to stretch. If the lining of the penile arteries becomes impaired, it can decrease the stretching of the artery and decrease blood flow. Decreased blood flow in the penile arteries can cause problems obtaining an erection.

The study medication Nebivolol controls blood pressure by relaxing smooth muscle around the lining of the arteries, thereby improving stretch and blood flow.

The primary objective is to determine if treatment with nebivolol improves endothelial function and erectile function in men with pre-hypertension and stage 1 hypertension

70 men will be enrolled into the study. Half of the subjects will receive active medication and half will receive a placebo. All men will receive educational informational handouts about blood pressure and behavior modifications to improve blood pressure. The study will last for 3 months for each subject. The expected recruitment time is one year, with a 2 year study completion goal. Subjects will have approximately 5 study visits.

Subjects will have initial/final blood work, a Rigiscan test (a take home penile erection test), two EndoPat tests to assess endothelium function, 3 SphygmoCor tests to assess central blood pressure, 2 sexual health questionnaires at 2 visits. Vital signs will be monitored at each visit to assess safety and effectiveness of the study medication.

DETAILED DESCRIPTION:
Randomized double-blind placebo-controlled study of 70 non-smoking pre-hypertensive men (BP 120-139 / 80-89) or with newly diagnosed stage 1 hypertension (BP > 140 but < 159/ 90-99) with erectile dysfunction receiving nebivolol (5-20mg) or placebo, along with lifestyle modifications, daily for 3 months to titrate BP to 120/80 or less.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Males 25-65
* Male Patients with ED (IIEF-5 ) Score > 13 and < 21

  o If a subject is using PDE5's( phosphodiesterase type 5 inhibitors), there must be a two week washout of PDE5 use, then in two weeks without PDE5 use; 4 attempts at sexual activity and an IIEF score < 21 on at least 2 of the four efforts
* Treatment naïve patients with Pre-hypertension (BP 120-139/80-89) or
* Stage 1 hypertension (BP > 140 but < 159/ 90-99)
* Patients in a stable, monogamous relationship
* Patients are able to comprehend and satisfactorily comply with protocol requirements
* Eugonadal Men : Total Testosterone 300 ng/dL-1000 ng/dL or greater, as well as men who are eugonadal with treatment.
* Non-smoker

Exclusion Criteria:

* Men with concomitant Type 1 or Type 2 Diabetes Mellitus
* Normal RigiScan at Baseline
* Concomitant use of ACE/ ARB (angiotensin receptor blocker)/ Beta-blocking agents/CCB (calcium channel blocker) / alpha-blocker
* Concomitant use of PDE5'S
* Currently Smoking
* Meeting any exclusion criteria for beta blocker use as stated in the nebivolol package insert
* Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
* Patients with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
* Patients who are unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Primary objective is to determine if treatment with nebivolol improves endothelial function and erectile function in men with pre-hypertension and stage 1 hypertension. This will be assessed by change in IIEF-5 at baseline, 2 and 3 months | baseline, 2 and 3 months
  The evaluation of the effect of the study medication will be assessed with IIEF questionnaire. This will be assessed by change in IIEF-5.

SECONDARY OUTCOMES:
Change in Endopat score | Measurement at baseline, and 3 months
  EndoPat test measures Endothelial function
Change in SphygmoCor results | SphygmoCor Measured at Baseline, 2 and 3 months
  Sphygmocor will measure change in pulse wave velocity and central blood pressure
Change in SQOLM score | questionnaire administered at SphygmoCor Measured at Baseline, 2 and 3 months
  SQOLM is the Sexual Quality of Life Male questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Miner, MD, Principal Investigator — The Miriam Hospital, a Lifespan partner
Locations (3):
- United States (3):
  - University Medicine, Providence, Rhode Island
  - Miriam Cardiology, Providence, Rhode Island
  - The Miriam Hospital / The Men's Health Center, Providence, Rhode Island